CLINICAL TRIAL: NCT03790579
Title: Is There Any Effect of Maternal Dietary Acid Load During Pregnancy on Arising Gestational Diabetes Mellitus?
Brief Title: Dietary Acid Load During Pregnancy and Gestational Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, F. Gülhan Samur, Professor doctor, Hacettepe University
Other Study IDs: Hacettepe Nutrition
Record Dates: First submitted 2018-12-28; First posted 2018-12-31 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Diabetes, Gestational; Dietary Habits
Keywords: Gestational diabetes mellitus; Dietary acid load; Pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with gestational diabetes: We randomly selected the 40 pregnant women diagnosed GDM by two-step procedure based on Carpenter-Coustan criteria at this hospital. The diagnosis of GDM was confirmed if at least 2 of 4 glucose levels exceed based on Carpenter-Coustan criteria: fasting ≥ 95 mg/dL (5.3 mmol/L), 1 hour ≥ 180 mg/dL ( 10.0 mmol/L), 2 hour ≥ 155 mg/dL (8.6 mmol/L), and 3 hour ≥ 140 mg/dL (7.8 mmol/L).
- Healthy women: We also randomly selected 40 healthy pregnant with normal serum glucose levels ≤129 mg/dL (7.2 mmol/L) after GCT.

SUMMARY:
Dietary habits resembling Western style, rich in animal protein and poor in fruit and vegetables, increase the body acid load, a predictor of type 2 diabetes risk. Recently, the studies related to relationships between dietary acid load and insulin resistance has become a growing interest but there are only a few study conducted with gestational diabetes mellitus (GDM). Therefore, the aim of this study was to evaluate the potential relationship between dietary acid load in second trimester, blood lipid profiles and GDM.

DETAILED DESCRIPTION:
This cross-sectional study conducted with 40 women with GDM diagnosed with two-step 100g oral glucose tolerance test and 40 healthy women, aged 21-41 years, between weeks of 14-28 of pregnancy, who attended the Department of Obstetrics and Gynecology of Gulhane Training and Research Hospital. Participants with polycystic ovary syndrome, chronic diseases, pre-GDM, or multiple pregnancies were excluded. Sociodemographic information was recorded via questionnaire and anthropometrics of women were measured.

Blood samples were taken after an overnight fasting. Dietary information was obtained by mean intakes of a 3-day food records (2 weekdays and 1 weekend day) and analyzed via nutrition analysis software. According to the data obtained from software analysis, animal protein (g/day) to potassium (g/day) ratio (AP/K), potential renal acid load (PRAL; mEq/day) score and net endogenous acid production (NEAP; mEq/day) were calculated from established algorithms to estimate dietary acid load. All nutrients were age and energy- adjusted before being introduced into the equation and tertiles of the scores were used for statistical analysis. ANOVA, ANCOVA and Logistic regression test were used. The study plan was approved by the Hospital's Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy,
* Aged in 20-40 years,
* Gestational age 24-28 weeks,
* Non-history of acute or chronic diseases.

Exclusion Criteria:

* History of GDM,
* Type 1 and 2 diabetes mellitus,
* Preeclampsia,
* Polycystic ovary syndrome,
* Thyroid disease
* Parathyroid disease,
* Metabolic bone disease,
* Kidney disease,
* Abnormal liver function,
* Multiple pregnancy
* Extreme values of energy intake in their dietary records (<1500 and >4000 kkal).

Ages: 21 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: In this observational cross-sectional study, 40 women with GDM and 40 healthy pregnant between 21-41 years in age, in their 24-28th gestational week applied to Gulhane Education and Research Hospital were recruited. This study must recruit 40 women for each group to have 80% study power with 5% type I error level to detect a clinically significant difference.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-01-05 (Actual); Primary Completion 2014-09-05 (Actual); Study Completion 2014-10-05 (Actual)

PRIMARY OUTCOMES:
Dietary acid load | 24-28. weeks of pregnancy
  According to the data obtained from software analysis, animal protein (g/day) to potassium (g/day) ratio (AP/K), potential renal acid load (PRAL; mEq/day) score and net endogenous acid production (NEAP; mEq/day) were calculated from established algorithms to estimate dietary acid load.

CONTACTS AND LOCATIONS:
Overall Officials: Gülhan SAMUR, Professor, Principal Investigator — Hacettepe University; Gözde EDE, MSci, Study Chair — Mehmet Akif Ersoy University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Della Guardia L, Thomas MA, Cena H. Insulin Sensitivity and Glucose Homeostasis Can Be Influenced by Metabolic Acid Load. Nutrients. 2018 May 15;10(5):618. doi: 10.3390/nu10050618. PMID 29762478
- [Background] Jayedi A, Shab-Bidar S. Dietary acid load and risk of type 2 diabetes: A systematic review and dose-response meta-analysis of prospective observational studies. Clin Nutr ESPEN. 2018 Feb;23:10-18. doi: 10.1016/j.clnesp.2017.12.005. Epub 2017 Dec 23. PMID 29460782
- [Background] Williams RS, Kozan P, Samocha-Bonet D. The role of dietary acid load and mild metabolic acidosis in insulin resistance in humans. Biochimie. 2016 May;124:171-177. doi: 10.1016/j.biochi.2015.09.012. Epub 2015 Sep 10. PMID 26363101
- [Result] Gaede J, Nielsen T, Madsen ML, Toft U, Jorgensen T, Overvad K, Tjonneland A, Hansen T, Allin KH, Pedersen O. Population-based studies of relationships between dietary acidity load, insulin resistance and incident diabetes in Danes. Nutr J. 2018 Oct 6;17(1):91. doi: 10.1186/s12937-018-0395-1. PMID 30292239
- [Result] Saraf-Bank S, Tehrani H, Haghighatdoost F, Moosavian SP, Azadbakht L. The acidity of early pregnancy diet and risk of gestational diabetes mellitus. Clin Nutr. 2018 Dec;37(6 Pt A):2054-2059. doi: 10.1016/j.clnu.2017.09.020. Epub 2017 Oct 3. PMID 29054469
- [Result] Miki A, Hashimoto Y, Tanaka M, Kobayashi Y, Wada S, Kuwahata M, Kido Y, Yamazaki M, Fukui M. Urinary pH reflects dietary acid load in patients with type 2 diabetes. J Clin Biochem Nutr. 2017 Jul;61(1):74-77. doi: 10.3164/jcbn.16-118. Epub 2017 Jul 1. PMID 28751813
- [Result] Kiefte-de Jong JC, Li Y, Chen M, Curhan GC, Mattei J, Malik VS, Forman JP, Franco OH, Hu FB. Diet-dependent acid load and type 2 diabetes: pooled results from three prospective cohort studies. Diabetologia. 2017 Feb;60(2):270-279. doi: 10.1007/s00125-016-4153-7. Epub 2016 Nov 17. PMID 27858141
- [Result] Williams RS, Heilbronn LK, Chen DL, Coster AC, Greenfield JR, Samocha-Bonet D. Dietary acid load, metabolic acidosis and insulin resistance - Lessons from cross-sectional and overfeeding studies in humans. Clin Nutr. 2016 Oct;35(5):1084-90. doi: 10.1016/j.clnu.2015.08.002. Epub 2015 Aug 12. PMID 26299332
- [Result] Akter S, Eguchi M, Kuwahara K, Kochi T, Ito R, Kurotani K, Tsuruoka H, Nanri A, Kabe I, Mizoue T. High dietary acid load is associated with insulin resistance: The Furukawa Nutrition and Health Study. Clin Nutr. 2016 Apr;35(2):453-459. doi: 10.1016/j.clnu.2015.03.008. Epub 2015 Mar 27. PMID 25863769